CLINICAL TRIAL: NCT02537808
Title: A Non-interventional Study of Lenalidomide (Revlimid®) in Combination With Dexamethasone as First Line Therapy in Transplant-ineligible Patients With Multiple Myeloma
Brief Title: Non-interventional Study of Lenalidomide / Dexamethasone as First Line Therapy in Patients With Multiple Myeloma
Acronym: FIRST-NIS
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-12315
Record Dates: First submitted 2015-08-24; First posted 2015-09-02 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this non-interventional study is to explore the safety, effectiveness and quality of life of lenalidomide / dexamethasone as first line treatment for transplant-ineligible patients with multiple myeloma in a real life setting.

DETAILED DESCRIPTION:
The introduction of new drugs that can be differently combined with conventional chemotherapy or low-dose dexamethasone has changed substantially the treatment paradigm for patients with multiple myeloma. A variety of treatment options is now available for elderly patients. To compare the efficacy and safety of continuous lenalidomide in combination with low-dose dexamethasone (Rd) until progression vs. Rd for 18 cycles/72 weeks (Rd18) vs. melphalan, prednisone and thalidomide (MPT) for 12 cycles/72 weeks a multicenter, open-label phase III study (MM-020/IFM 07-01, FIRST trial) was performed in transplant ineligible patients.

After market approval of lenalidomide for previously untreated transplant-ineligible patients with multiple myeloma, the purpose of the FIRST-NIS is to evaluate the safety, effectiveness and quality of life of lenalidomide in combination with dexamethasone as first line treatment of multiple myeloma in a real life setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (2008 WHO classification) requiring treatment (as defined by IMWG)
* Indication for treatment as assessed by the treating physician
* Decision for first line combination therapy with lenalidomide and low-dose dexamethasone
* No previous systemic therapy for multiple myeloma
* Ineligibility for transplantation
* Aged 18 years or older
* Written informed consent signed
* The conditions of the risk management plan/pregnancy prevention program (refer to the SmPC Revlimid®) must be followed by female and male patients
* Other criteria according to the SmPC. Special warnings and precautions of the SmPC have to be considered by the treating physician

Exclusion Criteria:

* Pregnant or breast-feeding women
* Any objections or contraindications according to the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplant-ineligible patients with previously untreated, symptomatic multiple myeloma (as defined by IMWG criteria) and with an indication for medical treatment as assessed by the investigator.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 24 months | 24 months

SECONDARY OUTCOMES:
To assess Median Overall Survival (OS) | 84 month
To assess safety and tolerability via AE and SAE reporting | 24 months
  AE, SAE and ADR are documented in the eCRF and will be used for safety assessment.
To assess Quality of Life (EORTC QLQ-C30 and MY20 | 24 months
  QoL data will be collected at baseline, after 3, 6, 12, 18 and 24 months
To assess duration of hospitalisation periods | 24 months
  To estimate hospital resource utilization by documenting how much time (days/weeks) patients spend in the hospital during their treatment period.
Overall Response Rate | 24 months
Median Progression-free survival (PFS) | 84 months
Median Time to Progression (TTP) | 84 months
Median Time to Response (TTR) | 24 months
Duration of Response | 84 months
Reason for treatment discontinuation | 84 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Nückel, Professor, Principal Investigator — Hämatologisch-Onkologische Schwerpunktpraxis
Locations (1):
- Hämatologisch-Onkologische Schwerpunktpraxis, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No